CLINICAL TRIAL: NCT04089189
Title: A Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of IMP4297 Capsules in Subjects With Germline and/or Somatic BRCA1/2 Mutation Positive Advanced Ovarian Cancer With at Least 2 Prior Lines of Standard Systemic Therapy
Brief Title: Study of IMP4297 in Patients With BRCA1/2 Mutation Ovarian Cancer
Acronym: SABRINA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP4297-2018-CN01
Record Dates: First submitted 2019-09-03; First posted 2019-09-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — senaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMP4297 (Experimental): 100 subjects to receive IM4297 orally.
  Interventions: Drug: IMP4297

INTERVENTIONS:
Drug: IMP4297 — IMP4297 100mg PO QD

SUMMARY:
A phase II, multi-center, open-label, single-arm, non-randomized study to evaluate the efficacy, safety and tolerability of IMP4297 capsules in subjects with germline and/or somatic BRCA1/2 mutated advanced ovarian cancer in china

DETAILED DESCRIPTION:
A total of 100 subjects with germline and/or somatic BRCA1/2 mutated advanced ovarian cancer is planned to be enrolled to observe the efficacy, safety, tolerability and PK profile of IMP4297.

The primary objective is to assess ORR in subjects with germline and/or somatic BRCA1/2 mutated advanced ovarian cancer with at least 2 prior lines of standard systemic therapy treated with IMP4297 capsules by independent imaging according to RECIST v1.1. Subjects will be treated until there is evidence of disease progression or any other discontinuation criterion is met. Best supportive care will be provided to all subjects and will be decided by investigators if there are no other specific restrictions within the protocol.

Four to seven blood samples (approximately 2 mL/sample) are planned to be collected for each enrolled subject for the popPK and/or dose-response evaluation. Sample collection visits are planned on Cycle (C) 1 Day (D) 1, C1D15, C2D1, C3D1 and C4D1. The actual administration time, dose and blood collection time should be accurately recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have to sign ICF prior to study-related procedures.
2. Female subjects ≥ 18 years of age with histologically or cytologically confirmed advanced non-mucinous ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer;
3. Germline and/or somatic BRCA1/2 mutation confirmed by central laboratory;
4. Disease relapse or progression after no less than 2 prior lines of platinum-based chemotherapy
5. No disease relapse or progression (based on clinical, CA125 or imaging) within 6 calendar months after the last platinum-containing regimen;
6. At least one measurable lesion confirmed by independent central imaging according to the criteria of RECIST v1.1;
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 0-1 (refer to Appendix 1);
8. Expected survival time ≥ 12 weeks;
9. Subjects, of sexually active and childbearing potential, and their spouses have to use contraception during the study and 90 days after the last dose of investigational drug (refer to Appendix 6 for acceptable contraception)

Exclusion Criteria:

1. Inadequate hematopoiesis or organ function (corrective treatment with blood products ≤ 14 days prior to the first dose of investigational drug, e.g. transfusion, etc., is not allowed):

   Absolute neutrophil count (ANC) <1.5×109/L; Hemoglobin (HGB) <9 g/dL; Platelet (PLT) <100×109/L; Total bilirubin (TBIL) >1.5 × upper limit of normal (ULN); Aspartate transferase (AST) and/or alanine aminotransferase (ALT) >3×ULN, AST and/or ALT of subjects with liver metastases >5×ULN; Creatine (Cr) >1.5 × ULN; International normalized ratio (INR) >1.5×ULN, or activated Partial thromboplastin time (aPTT) >1.5×ULN, (INR only for subjects who have not received anticoagulant therapy);
2. Have a history of radiation therapy < 4 weeks prior to the first dose of investigational drug, or chemotherapy, biological therapy, endocrine therapy or small molecule targeted therapy before the first dose of investigational drug (subject whose washout period ≥ 5 half-lives from the first dose of investigational drug can be enrolled);
3. Have received strong CYP3A4 inhibitors or strong CYP3A4 inducers prior to the first dose of investigational drug (washout period from the first dose of investigational drug ≥ 5 half-lives is allowed) or require continued treatment with these drugs during the study (as described in Section 6.9.2 of the protocol; refer to Appendix 2 for common CYP3A4 strong inhibitors or CYP3A4 strong inducers)
4. Have not recovered to NCI CTCAE v4.03 ≤ grade 1 from the toxicity of previous anti-tumor treatment, except alopecia;
5. Have had treatment with drugs targeting poly-ADP-ribose polymerase (PARP);
6. Clinically significant active infection;
7. History of clinically significant liver disease, including active viral or other hepatitis, history of alcohol abuse or cirrhosis; except for subjects with previous viral hepatitis confirmed to be inactive by polymerase chain reaction (PCR) assay;
8. Human immunodeficiency virus (HIV) infection;
9. Have congestive heart failure graded classification II or above assessed by New York Heart Association (NYHA); history of myocardial infarction or unstable angina within 6 months before treatment; history of stroke or transient ischemic attack within 6 months before treatment;
10. Subjects with active or untreated central nervous system metastases; subjects with treated brain metastases can be enrolled if the following criteria is met:

    Have no imaging progression ≥ 4 weeks after the end of treatment; The treatment completed ≥ 28 days prior to the first dose of investigational drug; Have no need to receive treatment with systemic corticosteroids (> 10 mg/day prednisone or equivalent) ≤ 14 days prior to the first dose of investigational drug;
11. Pregnant or lactating women
12. Subjects who had intestinal obstruction within 12 weeks prior to the first dose of investigational drug;
13. History of other malignancy within 5 years prior to the first dose of investigational drug;
14. Have had major surgery within 4 weeks prior to the first dose of investigational drug;
15. Subjects, at the discretion of the investigator, with poor compliance or with any factors unsuitable for participation in this trial; subjects, at the discretion of the investigator, to be unsuitable for participation in this study due to any clinical or laboratory abnormality.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 2) Female subjects ≥ 18 years of age with histologically or cytologically confirmed advanced non-mucinous ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer
Enrollment: 93 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
ORR | From enroll until a new antitumor therapy, disease progression, subject's withdrawal of informed consent form (ICF) and/or death，whichever came first, assessed up to 24 months
  Disease response as determined by Overall Response Rate per RECIST Version 1.1

SECONDARY OUTCOMES:
DOR | From enroll until a new antitumor therapy, disease progression, subject's withdrawal of informed consent form (ICF) and/or death，whichever came first, assessed up to 24 months
  Disease response as determined by Duration of Response per RECIST Version 1.1
FPS | From enroll until a new antitumor therapy, disease progression, subject's withdrawal of informed consent form (ICF) and/or death，whichever came first, assessed up to 24 months
  Disease response as determined by Progression Free Survival per RECIST Version 1.1
DCR | From enroll until a new antitumor therapy, disease progression, subject's withdrawal of informed consent form (ICF) and/or death，whichever came first, assessed up to 24 months
  Disease response as determined by Disease Control Rate per RECIST Version 1.1
CBR | From enroll until a new antitumor therapy, disease progression, subject's withdrawal of informed consent form (ICF) and/or death，whichever came first, assessed up to 24 months
  Disease response as determined by Clinical Benefit Rate per RECIST Version 1.1
OS | From enroll until subject's withdrawal of informed consent form (ICF) and/or death，whichever came first, assessed up to 24 months
  Disease response as determined by overall survival
Incidence of Treatment-Emergent Adverse Events | from the day of first enrolled of study drugs up to 30 days after the last administration
  Treatment-Emergent Adverse Events assessed by the investigator according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaohua.Wu, Shanghai, China

IPD SHARING:
Plan to Share IPD: No